CLINICAL TRIAL: NCT04149288
Title: Olive Oil Polyphenols and Cardiovascular Health Biomarkers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1484263
Record Dates: First submitted 2019-09-30; First posted 2019-11-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Normal Weight; Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-polyphenol olive oil (Active Comparator): Participants will consume 40 mL of high-polyphenol olive oil each day at home for 2 weeks.
  Interventions: Dietary Supplement: High-polyphenol olive oil
- Low-polyphenol olive oil (Active Comparator): Participants will consume 40 mL of low-polyphenol olive oil each day at home for 2 weeks.
  Interventions: Dietary Supplement: Low-polyphenol olive oil

INTERVENTIONS:
Dietary Supplement: High-polyphenol olive oil — High-polyphenol olive oil will be provided to study participants to consume at home. Participants will be asked to consume 40 mL each day for 2 weeks.
  Arms: High-polyphenol olive oil
Dietary Supplement: Low-polyphenol olive oil — Low-polyphenol olive oil will be provided to study participants to consume at home. Participants will be asked to consume 40 mL each day for 2 weeks.
  Arms: Low-polyphenol olive oil

SUMMARY:
The purpose of this research is to investigate whether consuming two different kinds of olive oil will change risk factors related to cardiovascular disease, including levels of good and bad cholesterol, levels of inflammation, and levels of gene expression.

DETAILED DESCRIPTION:
The purpose of this research is to investigate whether consuming two different kinds of olive oil will change risk factors related to cardiovascular disease, including levels of good and bad cholesterol, levels of inflammation, and levels of gene expression. Healthy individuals aged 20-45 with a BMI over 20 kg/m2 are eligible to participate. The study involves 5 visits (1 initial screening and 4 study visits) and will last about 8 weeks. There is a 2-week run-in period before starting the study, followed by two diet intervention periods each lasting two weeks, separated by a two-week washout period.

Participation in this study will involve an initial two-week run in period to become accustomed to the study diet. After this two week period, participants will be randomly selected to start either a high-polyphenol olive oil (extra virgin olive oil) or a low-polyphenol olive oil (refined olive oil); participants will consume the other oil during the second dietary intervention period lasting 2 weeks. During each phase of the study, participants will be asked to come to the University of California, Davis campus after a 10-12 hour overnight fast. At each visit, body measurements will be taken, a serving of olive oil and bread will be eaten, and three urine and blood samples will be collected over the course of 4 hours. Each study visit will involve three blood draws by a trained nurse or phlebotomist.

During the 8 weeks of the study, all olive products such as olives, olive oil, and olive containing products will need to be avoided. The study will provide olive oil to be eaten at home for each intervention phase. Additionally, the investigators will ask that nuts and high-polyphenol foods (mostly fruits and vegetables) be avoided in the diet. Detailed food diaries will be filled out and brought to study visits.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male and female subjects within the range of 20-45 years of age and BMI range of 18.5-29.9 kg/m2 for the healthy weight/overweight group and ≥ 30 kg/m2 for the obese group will be recruited.

Exclusion Criteria:

* Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant or lactating women, women planning to become pregnant in the next two months and prisoners will be specifically excluded
* Documented chronic diseases including diabetes, thyroid disease, kidney disease, metabolic syndrome, active cancer, previous cardiovascular events, history of gastric bypass or other GI issues related to fat absorption
* History of dyslipidemia or abnormal blood glucose levels (total cholesterol >240 mg/dL, elevated fasting blood glucose levels >125 mg/dL)
* Allergy to olives, inability to tolerate gluten or multiple allergies/intolerances that would significantly limit food intake
* Smoker or living with a smoker, illicit drug use, consuming >1 alcoholic drink/day, vaporizer and/or electronic cigarette use
* Extreme dietary or exercise patterns
* Recent weight fluctuations (>10% in the last 6 months)
* Taking prescription lipid medications or supplements that may affect lipoprotein metabolism, >1 g of fish oil/day, antioxidant supplements, cannabidiol (CBD) oil
* Taking exogenous hormones (e.g. hormonal birth control)
* Poor venous access
* Unwillingness to comply with study protocol

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Assessing the influence of olive oil polyphenols on cholesterol efflux | Through study completion, an average of 8 weeks
  Cholesterol efflux will be measured by assessing changes in reverse cholesterol transport rate in separated serum at each study time point (baseline, 2 hour, 4 hour) using a commercially available assay kit at each of the 4 study visits.
Assessing the influence of olive oil polyphenols on cholesterol ester transfer protein activity (CETP) | Through study completion, an average of 8 weeks
  Changes in CETP activity will be measured at each study time point (baseline, 2 hour, 4 hour) in plasma at each of the 4 study visits. The isolated plasma will be co-incubated with donor and acceptor molecules using a commercially available assay kit.
Assessing the influence of olive oil polyphenols on circulating oxidized LDL | Through study completion, an average of 8 weeks
  Measure for changes in circulating levels of oxidized LDL in separated plasma at each study time point (baseline, 2 hour, 4 hour) using a commercially available ELISA kit; measured in units of U/L at each of the 4 study visits.
Assessing the influence of olive oil polyphenols on blood lipid measurements | Through study completion, an average of 8 weeks
  Measure for changes in the levels of HDL and LDL in separated plasma; measured in units of mg/dL. Blood will be assessed for the fasting (baseline) sample only at each of the 4 study visits.
Assessing the influence of olive oil polyphenols on paraoxonase-1 (PON-1) activity | Through study completion, an average of 8 weeks
  Measure for changes in PON-1 activity in separated plasma at each study time point (baseline, 2 hour, 4 hour) at each of the 4 study visits. Activity will be calculated based on linear rates of hydrolysis of phenyl acetate to phenol.
Assessing the influence of olive oil polyphenols on peripheral blood mononuclear cells (PBMC) using ex vivo stimulation assays | Through study completion, an average of 8 weeks
  Measurement of changes in PBMC derived cytokines as a marker of inflammation at each study time point (baseline, 2 hour, 4 hour) at each of the 4 study visits. Assessment will be based on an increase or decrease in concentration in pg/ml.

SECONDARY OUTCOMES:
Assessing the influence of olive oil polyphenols on gene expression in mirco RNA in PBMCs | Through study completion, an average of 8 weeks
  Measure level of gene expression in micro RNA from PBMCs at each study time point (baseline, 2 hour, 4 ) at each of the 4 study visits. Assessment will be based on fold change between study arms.

OTHER OUTCOMES:
Food record analysis | Through study completion, an average of 8 weeks
  Use a computer program to check for study dietary requirements. Subjects are to avoid olives and olive containing products during study protocol periods. This will be done using a subject self-recorded 3-day food record submitted to study personnel.
Anthropometric measurements | Through study completion, an average of 8 weeks
  Measure waist (cm) and hip circumference (cm) before the start of drawing blood on study day protocols.
Measure for changes in weight | Through study completion, an average of 8 weeks
  Measure weight (kg) before the start of drawing blood on study day protocols.
Measure for changes in blood pressure | Through study completion, an average of 8 weeks
  Measure blood pressure (mmHg) before the start of drawing blood on study day protocols.
Assessing the influence of olive oil polyphenols on circulating cytokines | Through study completion, an average of 8 weeks
  Measure circulating cytokines in separated plasma at each study time point (baseline, 2 hour, 4 hour) at each of the 4 study visits. Commercially available ELISA kits will be used: TNF-a, IL-6, IL-1B, MCP-1, and ET-1.
Assessing the influence of olive oil polyphenols on urine metabolites | Through study completion, an average of 8 weeks
  Metabolomics will be performed on urine to assess for study compliance of consumption of the polyphenol containing olive oil versus the low-polyphenol containing olive oil at each of the 4 study visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Center, Davis, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-olive-oil-polyphenols-molecules-in-plant-based-food-and-cardiovascular-health-273896/